CLINICAL TRIAL: NCT04366895
Title: 3D Printing/Additive Manufacturing of Single- Implant Overdentures. A Randomized Controlled Clinical Trial.
Brief Title: 3D -Printed Single Implant Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Dina ElAwady, lecturer of Prosthodontics (principal investigator), October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSA
Record Dates: First submitted 2020-04-21; First posted 2020-04-29 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Edentulous Mouth
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Experimental): Participants in control group (Group-A) received conventional manufactured implant overdenture
  Interventions: Other: conventional single implant overdenture
- intervention (Experimental): participants in intervention group (Group-B) received CAD-CAM manufactured implant overdenture.
  Interventions: Other: 3d printed single implant overdenture

INTERVENTIONS:
Other: conventional single implant overdenture — conventional manufactured implant overdenture
  Arms: control
Other: 3d printed single implant overdenture — CAD-CAM manufactured implant overdenture.
  Arms: intervention

SUMMARY:
A randomized clinical trial (RCT) was designed. The participants were randomly allocated into either of the two groups intervention or control group each of 14 participants. Participants in control group (Group-A) received conventional manufactured implant overdenture while participants in intervention group (Group-B) received CAD-CAM manufactured implant overdenture.

DETAILED DESCRIPTION:
Introduction: Mandibular single implant overdenture is a well-established treatment modality that address limited financial resources of patients and simultaneously enabled the management of conventional complete denture problems. CAD/CAM technology helped to mitigate the problems encountered with conventional fabrication techniques, which results in improved dentures fit and retention. Therefore, the aim of the current trial study was to evaluate whether overdentures fabricated using CAD/CAM printed technology exhibited improved patient satisfaction, denture retention, implant survival rate and decreased post-insertion maintenance or not compared to overdentures manufactured using conventional techniques.

Methods: A randomized clinical trial (RCT) was designed. The participants were randomly allocated into either of the two groups intervention or control group each of seven participants. Participants in control group (Group-A) received conventional manufactured implant overdenture while participants in intervention group (Group-B) received CAD-CAM manufactured implant overdenture.

ELIGIBILITY:
inclusion criteria

* the participant should be completely edentulous ranging in age from 35 to 75 years
* Angle's class I skeletal relationship
* normal facial symmetry
* adequate inter-arch space not less than 12mm
* should be a cooperative patient -

Exclusion Criteria:

* temporomandibular disorders
* uncontrolled diabetes
* bleeding disorders or anticoagulant therapy
* flabby tissues or sharp mandibular residual ridge
* neuromuscular disorders
* Angle's class II and III skeletal relationship.
* Patients who were heavy smokers
* chemotherapy or radiotherapy or with severe psychiatric disorders

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-08-21 (Actual)

PRIMARY OUTCOMES:
Implant survival | 1 year
  The implants were considered surviving if they were clinically stable, functioning without any mobility

SECONDARY OUTCOMES:
Survival rate of overdentures | 1 year
  urvival rate of overdentures: (calculated by Incidence of mid-line fracture)
maximum biting force (MBF) | 1 year
  MBF was achieved bilaterally using Flexiforce A 301® force sensor and Arduino microcontroller with a crystal displa

CONTACTS AND LOCATIONS:
Overall Officials: Dina Elawady, PHD, Principal Investigator — Lecturer
Locations (1):
- Msa Uni, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No